CLINICAL TRIAL: NCT06005103
Title: Active Versus Sham Transcranial Pulsed Electromagnetic Field Headband Treatment for Major Depression: a Study Protocol for a Double-blinded Randomized Trial
Brief Title: A Randomized Clinical Trial Comparing Active Versus Sham T-PEMF Headband Treatment for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual); Danish Medical Association (Other); Doctor Gerhard Linds scholarship (Unknown); MoodHeadBand Aps (Unknown)
Responsible Party: Principal Investigator, Martin Balslev Jørgensen, Professor, dr. med., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2215332
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Moderate Depression; Severe Depressive Episode Without Psychotic Symptoms; Recurrent Depressive Disorder, Current Episode Moderate; Recurrent Depressive Disorder, Current Episode Severe Without Psychotic Symptoms
Keywords: Randomized Controlled Trial; Depression; Transcranial Pulsed Electro-Magnetic Fields (T-PEMF); Psychiatry; Cognition; Sleep
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients will receive either active (A) or placebo (B) treatment with the T-PEMF technology using af headband designed for this. The headbands will be chosen randomly from a bag containing a mix of headbands applying either treatment A or B. There will be two bags to choose from, one bag is designated for patients who use antidepressant drugs, the other is designated for patients who do not use antidepressant drugs at the time of inclusion in the study. The firm MoodHeadBand Aps was in control of the randomization procedure, making sure that each bag contained the same amount of headbands applying treatment A and B. An independent person tests the devices to ensure the devices function properly and to ensure that each bag contain an equal amount of active and placebo devices.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients and the research team don't know which headbands apply treatment A or B. The firm MoodHeadBand Aps was in charge of the randomization procedure, but will not know which patient receive treatment A or B. The headbands, control boxes and powerbanks are identifical. No difference can be seen or felt when the headbands are plugged into the control boxes and powerbanks. A small bulb will be lit when the controlbox is connected to a charged powerbank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (A) Patients diagnosed with moderate to severe depression without psychotic symptoms (Experimental): In total, 48 patients will be allocated to this arm.
  (In total, 117 patients will be included in the study. Data for the initial 21 patients included in the study could not be used to assess the antidepressant effect, why an increased number of participants was needed to secure the power for the trial. The technical difficulties have been addressed)
  Interventions: Device: Treatment with MoodHeadBand (T-PEMF treatment)
- (B) Patients diagnosed with moderate to severe depression without psychotic symptoms (Sham Comparator): In total, 48 patients will be allocated to this arm.
  (In total, 117 patients will be included in the study. Data for the initial 21 patients included in the study could not be used to assess the antidepressant effect, why an increased number of participants was needed to secure the power for the trial. The technical difficulties have been addressed)
  Interventions: Device: Inactive treatment with MoodHeadBand (Placebo)

INTERVENTIONS:
Device: Treatment with MoodHeadBand (T-PEMF treatment) — The patients will receive treatment with T-PEMF using a headband containing 20 coils placed symmetrically around the head of the patient. The device delivers 55 Hz magnetic field. Duration of treatment is 30 minutes once a day for 8 weeks.
  Arms: (A) Patients diagnosed with moderate to severe depression without psychotic symptoms
Device: Inactive treatment with MoodHeadBand (Placebo) — Patients will use an identical device, which does not deliver T-PEMF treatment. The patients will use the headband as the active group for 30 minutes, once a day, for 8 weeks.
  Arms: (B) Patients diagnosed with moderate to severe depression without psychotic symptoms

SUMMARY:
An 8-week, two-armed, randomized-controlled trial that examines the antidepressant effect of treatment with transcranial pulsed electromagnetic fields (T-PEMF) in patients diagnosed with moderate to severe depression using using a new device, the MoodHeadBand (MHB).

The participants will use an active or placebo MHB for 30 minutes daily for 8 weeks.

Additionally, the following research questions will be answered:

1. If there is a positive effect on the patients' emotional and non-emotional cognition after 8 weeks of active treatment compared to the sham group and if possible early changes in the emotional cognition can predict the treatment response after 8 weeks of treatment.

1. If the T-PEMF treatment provides improvement in restorative sleep after 8 weeks of treatment

DETAILED DESCRIPTION:
The purpose of this study is to clarify whether daily treatment over eight weeks with weak pulsating electromagnetic fields (T-PEMF) can achieve a safe effect on depression compared to the same treatment with a placebo T-PEMF. The study will furthermore explore possible effects on cognition and the hypothesized sleep-ameliorating effect of T-PEMF. Previous Danish studies have shown a significant antidepressant effect of other T-PEMF devices in the treatment of patients with depression.

The study is designed as a blinded, randomized study where active treatment is compared with inactive (placebo) treatment. At the same time, possible side effects in the use of the headband (MoodHeadBand, MHB) are investigated.

The project was initiated June 2024. Patients consecutively referred are asked after an initial interview whether they wish to participate in the study. If they give informed consent to this, they will be randomized to active or placebo treatment. The treatment itself takes place at home, 30 minutes once a day, for 8 weeks. "Treatment as usual" takes place in parallel to the study treatment, and consists of psychotherapy in a group or individually and antidepressive medications. Follow-ups will be conducted weekly either as visits at the clinic, via videocall or as telephone calls. The participants will receive weekly surveys they are encouraged to fill out prior to the weekly follow-ups. The severity of the depression, including its symptomatology will be examined weekly during the study, the cognitive test-battery is applied at baseline, week 1 and at the final visit, the patients sleep-pattern and possible disturbances are examined via the weekly surverys.

No significant side effects have been registered when using the same type of electromagnetic field treatment in the previous Danish studies. It has also been shown that it is possible to carry out the treatment at home without significant problems.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for moderate to severe depressive episode without psychotic symptoms according to the International Classification of Diseases and Related Health Problems 10th Revision (ICD-10)(The ICD-10 Classification of Mental and Behavioural Disorders: Diagnostic Criteria for Research 1993).
* Female participants: Females in the fertile age must deliver a negative pregnancy test, or previously have been sterilized.
* Female fertile participants: They must use safe contraceptive methods to be included in the study, and during the whole study.
* Has given written, informed consent to the trial.

Exclusion Criteria:

* Inability to speak or understand the Danish language.
* A current high risk of suicide (a score of 2 or more on the HAM-D-17 item 3).
* A co-morbid substance dependence.
* Bipolar affective disorder.
* Psychotic illness.
* Dementia.
* Other diagnoses of organic brain disease.
* The participant has any kind of implant, e.g. pacemakers or cochlear implants.
* Female participants: Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) | 8 weeks
  The IDS-SR is a 30-item self-report scale for measuring depressive symptoms, with satisfying psychometric features and good correlations with Hamilton-D17 (HAM-D17).

SECONDARY OUTCOMES:
Hamilton-D17 (HAM-D17) | 8 weeks
  A scale measuring depressive symptoms. Will be applied at baseline and at the end point
Hamilton-D6 (HAM-D6) | 8 weeks
  A scale measuring depressive symptoms. Will be applied at baseline and at the end point.
Quick Inventory of Depressive Symptomatology | 8 weeks
  A quick-version of the IDS questionnaire, that consists of 16 questions. Patients fill this assesment on a weekly basis during the study.
WHO-5 | 8 weeks
  This Well-Being Index consists of five items that are scored on a frequency response scale from "none of the time" (0) to "all of the time" (5).
Facial Expression and Recognition Test (FERT) | 8 weeks
  A test that assesses the patients recognition of - and attention to facial expressions as a part of the cognitive test battery that explores the patients "hot" cognition.
Emotional Categorization and Memory Test (ECMT) | 8 weeks
  A test that assesses the patient' self-referential memory with emotion laded words as a part of the cognitive test battery that explores the patients' "hot" cognition.
Screening of cognitive impairment in Psychiatry (SCIP) | 8 weeks
  A screening tool used to assess cognitive performance in psychiatric patients. The test includes List learning, delayed list learning, verbal fluency, visuomotor tracking tests. Explores the patients' "cold" cognitive mechanisms.
Trail Making Test B (TMT-B) | 8 weeks
  A test that assesses the patients' visual attention and ability to switch tasks. Explores the patients' "cold" cognitive mechanisms.
Sleep diary | 8 weeks
  The diary explores the patients sleep pattern and quality of sleep.
Udvalget for Kliniske Undersøgelser scale (UKU-24) | 8 weeks
  Side effects are assessed by the UKU-24 scale, including free text comments. Side effects will be assesed at week 1, 2, 4, 6 and at the end point.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Jørgensen, MD MSc, Principal Investigator — Psychiatric Center Copenhagen
Locations (1):
- Psychiatric Center Copenhagen, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
It is not possible to share individual participant data due to GDPR. Anonymised data after publishing might be available per request.

REFERENCES:
- [Derived] Brandborg Sorensen N, Haahr U, Larsen MP, Hansen J, Nyholm S, Videbech P, Bohr T, Miskowiak KW, Martiny K, Jorgensen MB. Active versus sham transcranial pulsed electromagnetic field headband treatment for major depression: protocol for a double-blinded randomised trial. BMJ Open. 2025 Oct 20;15(10):e104474. doi: 10.1136/bmjopen-2025-104474. PMID 41120157